CLINICAL TRIAL: NCT00296348
Title: An Open, Randomised, Multicentre Clinical Study to Investigate the Safety and Efficacy of Steroid Withdrawal With Tacrolimus, Mycophenolate Mofetil and Daclizumab Against Tacrolimus, Mycophenolate Mofetil and Steroids in Children After Kidney Transplantation
Brief Title: Comparing Efficacy and Safety of Steroid Withdrawal With Tacrolimus and MMF With Induction in Children After Kidney Transplantation
Acronym: TWIST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FG-506-02-43; PRG-EC-0243 (Other: Astellas Pharma Europe Ltd.)
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Kidney Transplantation
Keywords: Tacrolimus; Kidney Transplantation; Child; Treatment Outcome; Immunosuppression
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid; Daclizumab; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: tacrolimus; Drug: mycophenolate mofetil; Drug: steroids
- 2 (Experimental)
  Interventions: Drug: tacrolimus; Drug: mycophenolate mofetil; Drug: daclizumab

INTERVENTIONS:
Drug: tacrolimus — immunosuppression
  Other Names: Prograf; FK506
Drug: mycophenolate mofetil — oral
  Other Names: MMF
Drug: daclizumab — oral
  Arms: 2
Drug: steroids — oral
  Arms: 1

SUMMARY:
The primary objective of this study is to investigate the impact of early corticosteroid withdrawal in paediatric renal transplant patients on growth expressed as change in height standard deviation score (SDS) from baseline to end of study as the primary endpoint. The expected advantages are reduced growth suppression, lower incidence of arterial hypertension and post transplant diabetes mellitus (PTDM) and improved lipid metabolism, expressed by lower serum lipid values.

DETAILED DESCRIPTION:
Comparing efficacy & safety of steroid withdrawal with tacrolimus, mycophenolate mofetil (MMF) with induction in children after kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient younger than 18 but not younger than 2 years of age
* Skeletal age of boys < or = 17, girls < or = 15 years
* Patient has end stage kidney disease
* Female patient of childbearing potential must have a negative serum pregnancy test prior to enrolment and must agree to practice effective birth control during the study and 6 weeks thereafter.
* The patient, or in case the patient is a minor, the patient's parent(s) or their legal representative, has been fully informed and has given written informed consent

Exclusion Criteria:

* Patient has a most recently measured panel reactive antibody (PRA) grade of > or = 50%
* Patient is allergic to or intolerant of study medication
* Patient and/or donor is known to be HIV positive.
* Patient has significant liver disease
* Patient with malignancy or history of malignancy
* Patient has previously received or is receiving an organ transplant other than kidney.
* Patient has been previously enrolled in this study.
* Patient with the relapsing and non-diarrhoeal form of haemolytic uraemic syndrome.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 198 (Actual)
Dates: Start 2005-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Growth, expressed as change in height SDS from baseline to end of study is chosen as the primary endpoint. | 6 months

SECONDARY OUTCOMES:
Acute rejection: Incidence of and time to first biopsy proven acute rejection; overall frequency of acute rejections episodes; incidence of and time to first corticosteroid-resistant rejection; severity of biopsy-proven acute rejections (Banff97 criteria | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Physician, Study Director — Astellas Pharma Europe B.V.
Locations (34):
- Belgium (2):
  - Brussels
  - Leuven
- Prague, Czechia
- France (3):
  - Lyon
  - Nantes
  - Paris
- Germany (4):
  - Berlin
  - Cologne
  - Hanover
  - Heidelberg
- Budapest, Hungary
- Petah Tikva, Israel
- Italy (5):
  - Genova
  - Milan
  - Padua
  - Rome
  - Torino
- Warsaw, Poland
- Cluj-Napoca, Romania
- South Africa (2):
  - Cape Town
  - Johannesburg
- Gothenburg, Sweden
- Taipei, Taiwan
- Turkey (Türkiye) (2):
  - Ankara
  - Izmir
- United Kingdom (9):
  - Birmingham
  - Bristol
  - Glasgow
  - Leeds
  - Liverpool
  - London
  - Manchester
  - Newcastle upon Tyne
  - Nottingham

REFERENCES:
- See also: Link to FDA website — http://www.accessdata.fda.gov/scripts/cder/drugsatfda
- See also: Link to Results on EudraCT — https://www.clinicaltrialsregister.eu/ctr-search/trial/2005-001348-22/results